CLINICAL TRIAL: NCT00177879
Title: Schizophrenia Website Usability
Brief Title: Usability of a Website for People With Schizophrenia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was never granted for this study. No participants were ever enrolled.
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: University of Pittsburgh (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 0411096
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2008-08

CONDITIONS: Cognitive Deficits Related to Internet Use
Keywords: website; comparison

INTERVENTIONS:
Behavioral: website comparison

SUMMARY:
This study will determine the usability of a website for people with schizophrenia versus other websites designed for the same purpose.

DETAILED DESCRIPTION:
The objective of this study is to test and compare the usability of a website developed as part of a NIMH-funded project (see IRB #0208128), versus four other online websites in a effort to continue to improve website design elements and maximize usability by those identified with schizophrenia, a disease that produces cognitive impairments.

Prior usability testing done to evaluate a website developed as part of a NIMH-funded project (see IRB #0208128) was used to develop a website designed specifically to meet the needs of those with cognitive deficits. Generally, the website was well received. However, an implicit component of this project was to make quantitative statements comparing the website developed in this project to other existing websites for individuals with schizophrenia, in order to maintain and improve the usability of the website. As such, it is important to test the usability of this website versus other websites to continue to improve design elements and ease of use for those with serious mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia

Exclusion Criteria:

-

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Subject task performance data will be analyzed to determine what website properties influenced subject's performance of various assigned website search-related tasks.

SECONDARY OUTCOMES:
Website properties, such as reading level, font size, and amount of content on the homepage, etc will be used to determine what factors influence subject's performance, and thus the usability of the various websites.

CONTACTS AND LOCATIONS:
Overall Officials: Armando J Rotondi, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States